CLINICAL TRIAL: NCT02170077
Title: A Placebo-controlled Study to Investigate Safety and Efficacy of BIA 2-093 in Controlling Refractory Partial Seizures When Added to Ongoing Therapy
Brief Title: A Placebo-controlled Study to Investigate Safety and Efficacy of BIA 2-093
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-201
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Epilepsy
Keywords: Epilepsy; BIA 2-093
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ODG - once-daily group (Experimental): BIA 2-093 once-daily; Daily doses of BIA 2-093 were increased at four-weekly periods (400 mg, 800 mg and 1200 mg).
  Interventions: Drug: BIA 2-093
- TDG - twice-daily group (Experimental): BIA 2-093 twice-daily; Daily doses of BIA 2-093 were increased at four-weekly periods (400 mg, 800 mg and 1200 mg).
  Interventions: Drug: BIA 2-093
- PLG - placebo group (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIA 2-093 — BIA 2-093 (tablets) administered at increasing daily doses of 400 mg, 800 mg and 1200 mg once-daily or twice-daily, oral route
  Arms: ODG - once-daily group; TDG - twice-daily group
Drug: Placebo — Placebo tablets administered orally
  Arms: PLG - placebo group

SUMMARY:
The purpose of this study is to determine the efficacy of BIA 2 093 in the treatment of epileptic patients with refractory simple or complex partial seizures with or without secondary generalization.

DETAILED DESCRIPTION:
This clinical trial was performed as a multicentre, add-on, double-blind, randomised, placebo-controlled, phase II study. During the double-blind treatment phase (12 weeks) patients were assigned to three treatment groups receiving BIA 2 093 once daily (ODG - once-daily group), BIA 2 093 twice daily (TDG - twice-daily group) or placebo (PLG - placebo group), respectively. Daily doses of BIA 2 093 were increased at four-weekly periods (400 mg, 800 mg and 1200 mg).

On completion of the 12-week double-blind treatment period, a 1-week tapering period was scheduled.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18-65 years
* Patients with simple or complex partial seizures with or without secondary generalization since at least one year prior to randomisation visit
* At least 4 seizures per month within the last 2 months prior to randomisation
* Stable dose regimen of a maximum of two of the following AEDs: phenytoin, valproate, primidone, phenobarbital, lamotrigine, gabapentin, topiramate, clonazepam, during 2 months prior to randomisation
* Electroencephalogram (EEG) findings not contradicting the epilepsy diagnosis (e.g., primarily generalized epilepsy)
* Written informed consent.

Exclusion Criteria:

* Patient with nervus vagus stimulation
* Patient with primarily generalized seizures
* Known progressive neurological disturbance
* A history of status epilepticus within the past 3 months
* Seizure of non-epileptic origin
* Restricted legal competence and incapability to follow trial instructions
* Major psychiatric disorders
* Concurrent drug therapy with monoamine oxidase inhibitors or calcium channel blockers
* Need of excluded concomitant medication (see section 9.4.6.2)
* Use of oxcarbazepine or carbamazepine during the last 6 months before the randomisation visit
* Known hypersensitivity to oxcarbazepine or carbamazepine, or its metabolites
* Abuse of alcohol, drugs or medications
* History of relevant cardiac, renal, hepatic, endocrine, gastrointestinal, metabolic, hematologic or oncology disorders
* Second- or third-degree atrioventricular block not corrected with a pacemaker
* Relevant laboratory abnormalities (e.g., Na+< 130 mmol/L, alanine (ALT) or aspartate (AST) transaminase >2.0 times the upper limit of normal, white blood cell (WBC) count <3000 cells/mm3)
* Pregnancy, nursing or inadequate contraception in women of childbearing age (oral contraception should be combined with a barrier method)
* Participation in other clinical trials within the last 2 months
* History of non-compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2002-04; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BIAL - Portela & Cª, S.A., S. Mamede Do Coronado, S. Mamede Do Coronado, Portugal

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ODG - Once-daily Group | TDG - Twice-daily Group | PLG - Placebo Group
Started | 50 | 47 | 47
Intent to Treat (ITT) Population | 50 | 46 | 47
Completed | 41 | 34 | 35
Not Completed | 9 | 13 | 12
Not completed — Withdrawal by Subject | 3 | 4 | 2
Not completed — Adverse Event | 4 | 4 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Exclusion criteria | 2 | 2 | 5
Not completed — Exacerbation of seizures | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ODG - Once-daily Group | TDG - Twice-daily Group | PLG - Placebo Group | Total
Number analyzed (Participants) | 50 | 47 | 47 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (11.4) | 39.8 (11.9) | 40.4 (10.8) | 39.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 27 | 87
  Male | 21 | 16 | 20 | 57

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a 50% or Greater Reduction in Seizure Frequency (Further Referred to as "Responders") in a Treatment Period Compared to the Baseline Period
Time Frame: baseline, week 12
Measure: Number; unit: percentage of responders
Groups:
- ODG - Once Daily Group; TDG - Twice Daily Group; PLG - Placebo Group: Intent to treat (TT) Population
Arm/Group | ODG - Once Daily Group | TDG - Twice Daily Group | PLG - Placebo Group
Number analyzed (Participants) | 50 | 46 | 47
percentage of responders | 54 | 41 | 28

ADVERSE EVENTS:
Arm/Group | ODG - Once Daily Group | TDG - Twice Daily Group | PLG - Placebo Group
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/46 | 1/47
Other Adverse Events (participants affected / at risk) | 18/50 | 19/46 | 21/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ODG - Once Daily Group (N=50) | TDG - Twice Daily Group (N=46) | PLG - Placebo Group (N=47)
BACTERIAL INFECTION OF INTESTINES (Infections and infestations) | 1 | 0 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 1 | 0 | 0
VIRAL GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ODG - Once Daily Group (N=50) | TDG - Twice Daily Group (N=46) | PLG - Placebo Group (N=47)
Ear buzzing (Ear and labyrinth disorders) | 0 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 0
Diplopia (Eye disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0
Gastric pain (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 3 | 2
Vomiting (Gastrointestinal disorders) | 0 | 5 | 1
Chest pain (General disorders) | 0 | 1 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 1 | 0 | 1
Body temperature increased (Investigations) | 1 | 0 | 1
Creatine kinase increased (Investigations) | 0 | 0 | 3
Concentration impaired (Nervous system disorders) | 1 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 5 | 1
Drowsiness (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 8 | 3
Incoordination (Nervous system disorders) | 1 | 1 | 0
Somnolence (Nervous system disorders) | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Hair loss (Skin and subcutaneous tissue disorders) | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other